CLINICAL TRIAL: NCT01236469
Title: CryoValve® SG Aortic Human Heart Valve Combination Retrospective/Prospective, Multi-Center, Cohort Study
Brief Title: CryoValve® SG Aortic Human Heart Valve Combination Study
Acronym: SGAV
Status: Completed | Type: Observational
Sponsor: CryoLife, Inc. (Industry)
Responsible Party: Sponsor
Organization: CryoLife (Unknown)
Other Study IDs: SGA0903.000 - C(09/09)
Record Dates: First submitted 2010-10-01; First posted 2010-11-08 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Aortic Valve Stenosis; Aortic Valve Insufficiency
Keywords: Aortic Valve
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Retrospective Patients: Pediatric (21 years of age or younger) patients who received a CryoValve SG Aortic Valve distributed during the 2000 to 2003 period as an aortic valve replacement.
  Interventions: Procedure: Echocardiogram

INTERVENTIONS:
Procedure: Echocardiogram — A prospective follow-up Study Echocardiogram will be performed, as applicable, for those subjects who do not have echo data as of January 1, 2009.

SUMMARY:
The purpose of this study is to assess the probable benefit of CryoValve SG Aortic Human Heart Valve used in pediatric patients as an aortic valve replacement.

DETAILED DESCRIPTION:
The CryoValve SG aortic human heart valve is recovered from deceased human donors, treated with the SynerGraft® (SG) process,which is designed to reduce the donor cells present on the graft. The valve is then cryopreserved for storage until use. Removing cells from the heart valve has been shown to reduce a component of the immune response after implant compared to a standard allograft valve. However, it is not known how this affects the long-term durability of the valve.

ELIGIBILITY:
Inclusion Criteria:

* Patients implanted with a CryoValve SGAV as an aortic valve replacement.
* Patients who were ≤ 21 years of age at the time of implant.

Exclusion Criteria:

* Patients in whom the CryoValve SGAV was used as a patch or a non-valved conduit.
* Patients implanted with a CryoValve SGAV as a pulmonary valve replacement.
* Patients that were ≥ 22 years of age at the time of implant.

Ages: 6 Years to 27 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric (21 years of age or younger) patients who received a CryoValve SG Aortic Valve distributed during the 2000 to 2003 period as an aortic valve replacement.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2010-06; Primary Completion 2011-05 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Hemodynamic Performance | From Implant until Study Enrollment (on average, 7 years)
  Peak Aortic Gradient (or Peak Velocity), Mean Aortic Gradient, Aortic Insufficiency, Effective Orifice Area
Number of Adverse Events as a Measure of Safety | From Implant until Study Enrollment (on average, 7 years)
  Safety parameters will follow the guidelines for reporting morbidity and mortality after cardiac valvular operations as established by The American Association for Thoracic Surgery and The Society of Thoracic Surgeons.
  Evaluation of the following adverse events:
  * Mortality (all cause and valve-related)
  * Reoperation/reintervention
  * Explant
  * Endocarditis (all and valvular)
  * Thrombosis
  * Thromboembolism
  * Non-structural dysfunction
  * Perivalvular leak (all and major)
  * Bleeding (all and major)
  * Hemolysis
  * Calcification
  * Conduit failure

CONTACTS AND LOCATIONS:
Overall Officials: Scott B Capps, MS, Study Director — CryoLife, Inc.
Locations (9):
- United States (9):
  - Arizona Pediatric Cardiology Consultants, Phoenix, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Rady Children's Hospital, San Diego, California
  - The Children's Hsopital, Aurora, Colorado
  - Indiana University, Indianapolis, Indiana
  - C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - The Children's Mercy Hospital, Kansas City, Missouri
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma

REFERENCES:
- [Background] American College of Cardiology/American Heart Association Task Force on Practice Guidelines; Society of Cardiovascular Anesthesiologists; Society for Cardiovascular Angiography and Interventions; Society of Thoracic Surgeons; Bonow RO, Carabello BA, Kanu C, de Leon AC Jr, Faxon DP, Freed MD, Gaasch WH, Lytle BW, Nishimura RA, O'Gara PT, O'Rourke RA, Otto CM, Shah PM, Shanewise JS, Smith SC Jr, Jacobs AK, Adams CD, Anderson JL, Antman EM, Faxon DP, Fuster V, Halperin JL, Hiratzka LF, Hunt SA, Lytle BW, Nishimura R, Page RL, Riegel B. ACC/AHA 2006 guidelines for the management of patients with valvular heart disease: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (writing committee to revise the 1998 Guidelines for the Management of Patients With Valvular Heart Disease): developed in collaboration with the Society of Cardiovascular Anesthesiologists: endorsed by the Society for Cardiovascular Angiography and Interventions and the Society of Thoracic Surgeons. Circulation. 2006 Aug 1;114(5):e84-231. doi: 10.1161/CIRCULATIONAHA.106.176857. No abstract available. PMID 16880336
- [Background] Akins CW, Miller DC, Turina MI, Kouchoukos NT, Blackstone EH, Grunkemeier GL, Takkenberg JJ, David TE, Butchart EG, Adams DH, Shahian DM, Hagl S, Mayer JE, Lytle BW; Councils of the American Association for Thoracic Surgery; Society of Thoracic Surgeons; European Assoication for Cardio-Thoracic Surgery; Ad Hoc Liaison Committee for Standardizing Definitions of Prosthetic Heart Valve Morbidity. Guidelines for reporting mortality and morbidity after cardiac valve interventions. J Thorac Cardiovasc Surg. 2008 Apr;135(4):732-8. doi: 10.1016/j.jtcvs.2007.12.002. No abstract available. PMID 18374749
- [Background] Zehr KJ, Yagubyan M, Connolly HM, Nelson SM, Schaff HV. Aortic root replacement with a novel decellularized cryopreserved aortic homograft: postoperative immunoreactivity and early results. J Thorac Cardiovasc Surg. 2005 Oct;130(4):1010-5. doi: 10.1016/j.jtcvs.2005.03.044. PMID 16214512